CLINICAL TRIAL: NCT02113046
Title: Prospective Randomized Study to Decrease Pancreatic Fistula Rate
Brief Title: Pancreatic Stump Closure After Distal Pancreatic Resection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis does not show good results
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Anne Antila, MD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R09131
Record Dates: First submitted 2014-03-26; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Distal Pancreatic Resections
Keywords: pancreas; pancreatico-jejunal anastomosis; postoperative pancreatic fistulae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pancreatico-jejunal anastomosis (Active Comparator): patients in which the finnish binding pancreatico-jejunal anastomosis is techically possible to perfom during distal pancreatic resektion
  Interventions: Procedure: pancreatico-jejunal anastomosis
- traditional anastomosis (Active Comparator): pancreatic resections with traditional stump closure
  Interventions: Procedure: traditional anastomosis

INTERVENTIONS:
Procedure: pancreatico-jejunal anastomosis
  Arms: pancreatico-jejunal anastomosis
Procedure: traditional anastomosis
  Arms: traditional anastomosis

SUMMARY:
The aim of this study is to investigate whether finnish binding pancreatico-jejunal anastomosis is feasible and prevents the risk for post operative pancreatic fistula after distal pancreeatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patiens which the distal pancreatic resektions
* the type of resections that is techically possible with finnish binding panceatico-jejunal anastomosis

Exclusion Criteria:

* if the pancreas is not suitable for this kind of anastomosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
postoperative pancreatic fistula rata | 30 days

SECONDARY OUTCOMES:
Number of patients with resection margin on the left side of portal vein as a measure of feasibility. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University hospital, Tampere, Pirkanmaa, Finland